CLINICAL TRIAL: NCT06854094
Title: Consolidation Therapy with Immune Reconstitution Therapy (cladribine) in Relapsing Multiple Sclerosis Patients Following a Treatment with Anti-CD20 Compounds: a Pivotal Study
Brief Title: Consolidation Therapy with Cladribine in Relapsing Multiple Sclerosis Patients
Acronym: OCR_CLAD
Status: Recruiting | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: 3B Biotech Research (Other)
Responsible Party: Principal Investigator, Chiara Zecca, Prof. dr.ssa med., Ente Ospedaliero Cantonale, Bellinzona
Other Study IDs: OCR_CLAD INSI.SM.2403
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: Switch to Cladribine
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
To investigate the impact on IgG and IgM concentration, infection risk and effectiveness of switching from anti-CD20 to cladribine compared to continued anti-CD20 treatment over 2 years in relapsing MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing MS according to Lublin [23]

EDSS ≤7.0 - Male and female patients with age >18 years - Treatment with ocrelizumab or rituximab for ≥12 months and/or having received ≥ 1.2 / 1.0 gr, respectively - For CLAD_GROUP: Planning to switch to cladribine because of concerns about increased risk of infections related to long term anti-CD20 therapies, defined as at least 3 infectious events/year or a serious infection under anti-CD20 and/or a documented decrease of ≥ 5% IgG and/or a level of IgG below 7 gr/L compared to pre- anti-CD20 therapy (will be considered as CLAD_GROUP)

- For OCR_GROUP and RTX_GROUP: continuing anti-CD20 therapies (considered as OCR_GROUP and RTX_GROUP with ocrelizumab with rituximab treatment, respectively)

- Anti-CD20 and Cladribine are prescribed according to Swiss and European SmPC.

Exclusion Criteria:

* Non-relapsing MS

Pregnancy or lactation - Contraindication to receive cladribine or to continue anti-CD20 therapies according to local label - Inability to complete an MRI - Known presence of other neurological disorders which may mimic MS including but not limited to: neuromyelitis optica, Lyme disease, untreated vitamin B12 deficiency, neurosarcoidosis and cerebrovascular disorders - Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study

- Significant or uncontrolled somatic disease or any other significant disease that may preclude patient from participating in the study

- Known active bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds Infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit

- History of progressive multifocal leukoencephalopathy (PML)

- Active malignancy, including solid tumors and hematological malignancies, except basal cell carcinoma, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that have been previously completely excised with documented, clear margins

- History of alcohol or drug abuse within 24 weeks prior to baseline

- Lymphocyte count < 1000 /μL

- AST/SGOT or ALT/SGPT ≥ 3.0 Upper Limit of Normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruited population will consist in 70 patients with RMS treated with anti-CD20 (ocrelizumab or rituximab) for ≥12 months and/or having received 1.2/1.0 gr, respectively, of the previously mentioned drugs that are switched to cladribine because of concerns about increased risks of infections during long term anti-CD20 therapies (defined as at least 3 infectious events/year and/or a serious infection under anti-CD20 treatment and/or a documented decrease of ≥ 5% IgG compared to pre anti-CD20 therapy and/or a level of IgG below 7 gr/L (CLAD_GROUP)).
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
changes in IgG serum concentrations 6, 12, 24 months after switching to cladribine following a treatment with anti-CD20 therapies compared to the last 12 months of antiCD20 therapy, and to patients continuing anti-CD20. | From enrollment to the end of treatment at 24 months
  1. Explore the impact of switching from continuous anti-CD20 to cladribine on serum immunoglobulins and other clinical, imaging and biomarker parameters in a large, multicenter, international population of MS patients
  2. Extend the observation period to at least 2 years in order to see a stabilization or an improvement of immunoglobulin concentration and a related decreased infection rate in patients switching to cladribine compared to those continuing anti-CD20.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Lugano, Istituto di Neuroscienze Cliniche della Svizzera Italiana, Via Tesserete 46,, Lugano, Canton Ticino, Switzerland